CLINICAL TRIAL: NCT04170322
Title: Randomized Controlled Trial Comparing Introduction Time of Thin Pvc Versus Thick Silicone Gastric Calibration Tubes for Sleeve Gastrectomy.
Brief Title: Comparing Pvc or Silicone Gastric Calibration Tube During Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, Prof Dr, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019RCTgastrictube
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Surgery; Calibration Tube

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thin pvc gasrtric calibration tube (Experimental): thin pvc gastric calibration tube is inserted after intubation to release gas from the stomach, then moved in correct position to help surgeon construct a sleeve gastrectomy.
  Interventions: Device: thin pvc gastric tube
- thick silicone gastric calibration tube (Active Comparator): thick silicone gastrric calibration tube is inserted after intubation to release gas from the stomach, then moved in correct position to help surgeon construct a sleeve gastrectomy
  Interventions: Device: thick silicone gastric tube

INTERVENTIONS:
Device: thin pvc gastric tube — a thin pvc gastric tube of 40 Fr for sleeve is used to guide the surgeon
  Arms: thin pvc gasrtric calibration tube
Device: thick silicone gastric tube — a thick silicone gastric tube 40 Fr for sleeve is used to guide the surgeon
  Arms: thick silicone gastric calibration tube

SUMMARY:
Time from 40 Fr gastric calibration tube introduction on surgical request till first stapling is measured as introduction time.

Problems to advance are noted A note is made If change to other type of gastric tube is needed

DETAILED DESCRIPTION:
when ready to perform sleeve gastrectomy anesthesiologist is asked to introduce 40 Fr gastric calibration tube. A clock is running till first staple is fired as a measure of time to introduce.

If problems to position 40 Fr gastric calibration tube correctly, if resistance to advance, change to other type of gastric tube and check again difficulties. Make a note of problems and reason to change.

ELIGIBILITY:
Inclusion Criteria: only primary sleeve gastrectomy

-

Exclusion Criteria:

* revision procedure
* known eosophageal or gastric anatomical abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
introduction time | intraoperative
  time from introduction until first staple in minutes

SECONDARY OUTCOMES:
rate of changing tube | intraoperative
  Impossible for correct positioning requiring change to another tube

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paul Mulier, Principal Investigator — AZ Sint-Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium